CLINICAL TRIAL: NCT00905723
Title: Effects of Isoflavone and Estrogen in Sex Response in Climacteric Women
Brief Title: The Effects of Isoflavone and Estrogen in Sex Response in Climacteric Women
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Teresa Raquel Embiruçu de Araújo, Universidade Federal de São Paulo - Departamento de Ginecologia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0759/08
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Postmenopausal Symptoms
Keywords: climacterium; sexual life; isoflavone; estrogen; McCoy's sexual questionnaire; Kupperman index
MeSH Terms: interventions — Estradiol; Isoflavones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Estrogen (Experimental): Women randomized to this group will receive daily pills containing 1 mg of estradiol
  Interventions: Drug: estradiol
- Isoflavone (Experimental): Women randomized to this group will receive daily pills of 150 mg isoflavone
  Interventions: Drug: isoflavone
- Placebo (Placebo Comparator): Women randomized to this group will be administered daily placebo pills
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: estradiol — 1 mg daily for 6 months
  Arms: Estrogen
Drug: isoflavone — 150 mg isoflavone daily for 6 months
  Arms: Isoflavone
Drug: Placebo — sugar pill daily for six months
  Arms: Placebo

SUMMARY:
Climacterium is marked by hypoestrogenism and it is associated to drastic vasomotors symptoms, genital atrophy and humor alteration. Additionally, these symptoms impair sexual life and life quality. These effects can be counteracted by administration of estrogen therapy. However, estrogen therapy has side effects and isoflavone has been proposed as an estrogen substitute in reposition therapy. The aim of the randomized controlled trial is to evaluate the effects of isoflavone in the sex life assessed by a modified McCoy's sexual questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* women aged 45-65 years old
* presenting climacteric symptoms
* sexual complaints

Exclusion Criteria:

* hormonal therapy
* counter indication to hormonal therapy
* uncontrolled comorbidities

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
McCoy's sexual questionnaire | at recruitment and six months later

SECONDARY OUTCOMES:
Kupperman's index | at recruitment and six months later

CONTACTS AND LOCATIONS:
Overall Officials: Mauro A Aidar, M.D., PhD, Study Chair — Universidade Federal de São Paulo
Locations (1):
- Ambulatório de Ginecologia Endócrina, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Universidade Federal de São Paulo's web page — http://www.unifesp.br